CLINICAL TRIAL: NCT02771457
Title: Managing Infliximab Reinduction After Temporary Discontinuation of Drug
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-01180
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: Influximab; IFX; Remicade
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infliximab at weeks 0,2, and 6 (Experimental): In this arm subjects will receive re-induction treatment of infliximab at weeks 0,2, and 6.
  Interventions: Drug: Infliximab at weeks 0,2, and 6
- Infliximab at weeks 0,4, and 8 (Experimental): In this arm subjects will receive re-induction treatment of infliximab at weeks 0, 4, and 8
  Interventions: Drug: Infliximab at weeks 0,4, and 8
- Infliximab at weeks 0, and 8 (Active Comparator): In this arm subjects will not be randomized. They will receive re-induction therapy weeks 0 and 8.
  Interventions: Drug: Infliximab at weeks 0 and 8

INTERVENTIONS:
Drug: Infliximab at weeks 0,2, and 6
  Arms: Infliximab at weeks 0,2, and 6
Drug: Infliximab at weeks 0,4, and 8
  Arms: Infliximab at weeks 0,4, and 8
Drug: Infliximab at weeks 0 and 8 — For physicians who do not feel comfortable enrolling patients in a randomized trial of infliximab re-induction they will have the option of enrolling their patients in an arm that resumes maintenance therapy only instead at 0 and 8 weeks.
  Arms: Infliximab at weeks 0, and 8

SUMMARY:
The primary purpose of the project is to determine what is the best schedule for restarting infliximab in patients with inflammatory bowel disease (IBD) specifically ulcerative colitis and Crohn's disease, who have undergone infliximab infusions before. The primary endpoint would be the failure rate; the need to discontinue infliximab or change treatment. A secondary aim will be to determine if infliximab drug and antibody levels can predict clinical outcomes at 1 year. Other secondary outcomes include comparing short-term and long-term steroid free remission rate, and serum and fecal inflammatory markers in response to infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older who are willing and able to provide informed consent
* HIstory of IBD (Crohn's disease, ulcerative colitis, indeterminate colitis) by standard clinical, histological, and radiographic date.
* History of stable clinical response to prior IFX induction and regular maintenance dosing, as determine by enrolling clinician.
* Prior to drug holiday, was on stable dose of infliximab for at least 3 infusions at regular maintenance intervals
* Infliximab drug holiday for at least 12 weeks.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Pregnant patients
* Prior history of serious infusion reaction to IFX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Failure Rate | One year
  Defined by the number of patients who discontinued or are adjusting their dosage of Infliximab.

SECONDARY OUTCOMES:
Short-term clinical response | One year
  The physician will determine the presence or absence of IBD (Inflammatory Bowel Disease) using his clinical judgement based on clinical disease indices and serum inflammatory biomarkers.
Long-term clinical response | One year
  The physician will determine the presence or absence of IBD (Inflammatory Bowel Disease) using his clinical judgement based on clinical disease indices and serum inflammatory biomarkers.
Short-term changes in patient Quality of Life | One Year
  This will be measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
Long-term changes in patient Quality of Life | One Year
  This will be measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
Fecal calprotectin measurements | One year
  This will be measured by ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: Lea Chen, Principal Investigator — NYU Langone Health